CLINICAL TRIAL: NCT04920981
Title: Real World Effectiveness and Treatment Sequences in Patients With Extensive Stage SCLC Who Received Atezolizumab Combined With Chemotherapy as Part of the French Early Access Program (ATU).
Brief Title: Atezolizumab Combined With Chemotherapy in Extensive Stage SCLC
Acronym: CLINATEZO
Status: Completed | Type: Observational
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: Roche Pharma AG (Industry); GFPC (Unknown)
Responsible Party: Sponsor
Other Study IDs: IFCT-1905
Record Dates: First submitted 2021-04-28; First posted 2021-06-10 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; atezolizumab; IFCT; Real-world study
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: atezolizumab — observational

SUMMARY:
CLINATEZO cohort will evaluate overall survival, real world progression-free survival, best response and duration of treatment in patients with advanced, metastatic Small Cell Lung Cancer (SCLC) who received atezolizumab combined with chemotherapy part of the French Early Access Program (ATU). Subsequent treatments (treatment delivered immediately after treatment with atezolizumab and chemotherapy) will be recorded. Those outcomes will be correlated to clinical, pathological, and radiological characteristics of patients.

DETAILED DESCRIPTION:
Standard-of-care first-line treatment for advanced, metastatic Small Cell Lung Cancer is platinum chemotherapy (carboplatin or cisplatin) with etoposide. Despite response rates of 60 to 65%, limited progress has been made in more than two decades; outcomes remain poor, with a median overall survival of approximately 10 months. Small cell lung cancer has a high mutation burden, which suggests that these tumors may be immunogenic and could respond to immune-checkpoint inhibitors.

Atezolizumab is a humanized monoclonal anti-programmed death ligand 1 (PD-L1) antibody that inhibits PD-L1-programmed death 1 (PD-1) and PD-L1-B7-1 signaling and restores tumor-specific T-cell immunity.

The addition of atezolizumab to chemotherapy in the first-line treatment of advanced, metastatic Small Cell Lung Cancer has been granted access for patients in France part of an Early access program (ATU), in May 2019.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed extensive stage Small Cell Lung Cancer at time of initiation of treatment with atezolizumab and chemotherapy.
* Patients who were informed about the study and accepted for their data to be collected.
* Patients who received at least one dose of treatment with atezolizumab and chemotherapy as part of the French Early Access Program (ATU program) and have been accepted within this ATU program
* Selection period spans from May 6th 2019 until January 31st 2020 for initiation of treatment with atezolizumab and chemotherapy.

Exclusion Criteria:

* Patients enrolled in a clinical trial assessing treatment with a combination of atezolizumab and chemotherapy. (ATU was granted to patients unable to meet eligibility criteria for on-going recruiting trials, unable to participate to other clinical trials, or because other medical interventions were not considered appropriate or acceptable).
* Patients who were included in the French Early Access Program (ATU program) but did not receive any atezolizumab and chemotherapy treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed extensive stage Small Cell Lung Cancer at time of initiation of treatment with atezolizumab and chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 518 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | OS will be measured at 6 months, 12 months, 24 months, 3 years and 4 years.
  OS is defined as the time from the first dose of treatment with atezolizumab and chemotherapy to death from any cause.

SECONDARY OUTCOMES:
Pattern of tumor progression | Study completion (4 years)
  site of disease progression after treatment with atezolizumab and chemotherapy
Duration of treatment | Study completion (4 years)
  time from first dose of treatment to discontinuation of treatment (interruption of more than 2 months) with atezolizumab and/or chemotherapy
Presence of liver metastases | At atezolizumab initiation
  yes/no
Performance Status | At atezolizumab initiation
  score (0/1/2/3/4/5)
Real-world progression-free survival (rwPFS) | rwPFS will be measured at 6 months, 12 months, 24 months, 3 years and 4 years.
  rwPFS is defined as the time from first dose of treatment with atezolizumab and chemotherapy to first occurrence of disease progression or death from any cause during the study
Best response | Study completion (4 years)
  best response recorded from the start of treatment with atezolizumab and chemotherapy until disease progression or start of further anti-cancer treatment
Sex | At inclusion
  male/female
Age | At atezolizumab initiation
  years

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRARD, Principal Investigator — Paris - Institut Curie; Lionel FALCHERO, Principal Investigator — Chalon-sur-Saône - CH
Locations (2):
- France (2):
  - Chalon-sur-Saône - CH, Chalon-sur-Saône
  - Paris - Institut Curie, Paris

REFERENCES:
- See also: Article — https://pubmed.ncbi.nlm.nih.gov/37757576/